CLINICAL TRIAL: NCT07323745
Title: Long-Term Effects of Mobithron Advance on Knee Osteoarthritis
Brief Title: Long-Term Effects of Mobithron Advance on Knee Osteoarthritis Aims to Investigate the Effects of Mobithron Advance on OA Progression
Acronym: mobithron adv
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: BREGO Life Sciences Sdn Bhd (Unknown)
Responsible Party: Principal Investigator, Amran Ahmed Shokri, Professor, Universiti Sains Malaysia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mobithron grant
Record Dates: First submitted 2025-12-07; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis (OA) of the Knee
Keywords: Mobithron Advance
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This Mobithron study uses a prospective, single-arm interventional clinical trial model, where all patients will receive Mobithron Advance daily for 12 months. This design allows you to follow participants forward in time and directly assess the effects of the intervention on knee osteoarthritis outcomes, including cartilage preservation, pain reduction, functional improvement, and safety. The single-arm approach is suitable for an early-stage study of a novel therapeutic, focusing on generating essential safety and efficacy data before progressing to randomised controlled trials. By including patients across Kellgren-Lawrence grades 1-3, the study also explores how disease severity influences treatment response.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobithron Advance Arm (Experimental): Treatment Arm will receive one Mobithron Advance oral tablet daily for 12 months. Outcomes will be assessed include cartilage preservation (MRI), pain (VAS), function (WOMAC), and safety (renal function and adverse events)
  Interventions: Drug: Type 2 collagen

INTERVENTIONS:
Drug: Type 2 collagen — This study's intervention is undenatured type II collagen (UC-II) oral tablets, one daily for 12 months, targeting knee osteoarthritis (KL grade 1-3). It differs from other interventions such as glucosamine, chondroitin, hyaluronic acid, or NSAIDs by working through an oral tolerance mechanism with the potential to preserve cartilage and modify disease progression, rather than providing only short-term symptom relief.
  Other Names: Mobithron Advance

SUMMARY:
The goal of this clinical trial is to learn if the Mobithron Advance drug works to treat and slow the progression of osteoarthritis (OA) in patients. It will also learn about the safety and long-term effects of this drug. The main questions it aims to answer are:

* Does long-term administration of Mobithron Advance can modify the progression of knee osteoarthritis with Kellgren-Lawrence grade 1 to 3 in HUSM patients?
* Does long term usage of Mobithron Advance has safety profile? Researchers will compare the Mobithron Advance drug to a placebo (a look-alike substance that contains no drug) to see if said drug works to treat OA.

Participants will:

* Undergo pre-study assessment (baseline assessments) during first visit
* Take oral Mobithron Advance daily for 1 year
* Visit the clinic once at 3 months, 6 months and 12 months intervals from the initial visit for follow up assessments

DETAILED DESCRIPTION:
The study will be conducted as a prospective single-arm trial with a one-year follow-up at the Orthopaedic Clinic, Hospital Universiti Sains Malaysia (HUSM), Malaysia. Participants will include adults over 50 years old diagnosed with primary knee osteoarthritis (OA) of Kellgren-Lawrence grade 1 to 3, based on clinical and radiological criteria. A total of 84 patients will be recruited, accounting for a 10% dropout rate, and will receive daily oral Mobithron Advance for 12 months. Pain will be assessed monthly using the Visual Analogue Scale (VAS) and physical function will be evaluated with the WOMAC index at follow-up visits. Cartilage preservation will be measured through MRI scans at baseline, six months, and twelve months, using a cartilage-specific 3D WATSc sequence to monitor central femoral condyle thickness. Safety and tolerability will be assessed by monitoring renal function, including creatinine and eGFR, alongside recording any adverse events. Data will include demographics, clinical outcomes, and radiological findings, and will be analysed using descriptive statistics, paired t-tests or Wilcoxon signed-rank tests, and linear mixed-effects models to evaluate changes over time.

ELIGIBILITY:
Inclusion Criteria:

* Males and female patients above 50 years old at the time of recruitment.
* OA Diagnosis: Patients with one or both knee osteoarthritis according to clinical and radiological criteria of the American College of Rheumatology (ACR).
* OA Grade: Kellgren Lawrence grade 1-3

Exclusion Criteria:

* Secondary arthritis (e.g., rheumatoid arthritis, psoriatic arthritis).
* History of joint surgery.
* Patients who received steroid injection treatment within the last 3 months or hyaluronic acid injection treatment within the last 6 months.
* Contraindications to Mobithron Advance (e.g., known allergies, severe liver or kidney disease).
* Patients planning for knee surgery within the research period.
* Patients on pharmacological treatment for osteoarthritis, other than rescue analgesic agent, e.g: glucosamine, chondroitin, oral steroid

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
to assess the thickness of cartilage in osteoarthritic knee included in the study at 3 stages. pre treatment, mid treatment and post treatment. | 1 year
  in term of cartilage assessment, MAGNETIC RESONANCE IMAGING (MRI) PROTOCOL is going to be used; in which, Multiplanar reconstruction (MPR) of the 3D WATSc image will be done to determine the location of central medial femoral condyle cartilage, where thickness of the central medial femoral condyle (cMF) cartilage will be measured on sagittal plane at the most central weight bearing surface.
  with the above outcome measure, the study can look into Mobithron able to preserve and regenerate cartilages in patients, slowing and reversing cartilage losses as well as disease progression.

SECONDARY OUTCOMES:
assessment of pain score in knee osteoarthritic patient | 1 year
  The outcomes is measured using visual analogue score (VAS) for pain intensity assessment at 3 months interval

OTHER OUTCOMES:
functional assessment of patient with osteoarthritic knee included in this study | 1 year
  WOMAC osteoarthritis index is going to be used to assess the functionality of the patient with osteoarthritic knee included in the study, assessment is done every 3 months durint the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Univerisiti Sains Malaysia (HUSM), Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
to protect participant personal data

REFERENCES:
- [Background] Lugo JP, Saiyed ZM, Lau FC, Molina JP, Pakdaman MN, Shamie AN, Udani JK. Undenatured type II collagen (UC-II(R)) for joint support: a randomized, double-blind, placebo-controlled study in healthy volunteers. J Int Soc Sports Nutr. 2013 Oct 24;10(1):48. doi: 10.1186/1550-2783-10-48. PMID 24153020
- [Background] Kalman DS, Heimer M, Valdeon A, Schwartz H, Sheldon E. Effect of a natural extract of chicken combs with a high content of hyaluronic acid (Hyal-Joint) on pain relief and quality of life in subjects with knee osteoarthritis: a pilot randomized double-blind placebo-controlled trial. Nutr J. 2008 Jan 21;7:3. doi: 10.1186/1475-2891-7-3. PMID 18208600
- [Background] Crowley DC, Lau FC, Sharma P, Evans M, Guthrie N, Bagchi M, Bagchi D, Dey DK, Raychaudhuri SP. Safety and efficacy of undenatured type II collagen in the treatment of osteoarthritis of the knee: a clinical trial. Int J Med Sci. 2009 Oct 9;6(6):312-21. doi: 10.7150/ijms.6.312. PMID 19847319
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19847319/